CLINICAL TRIAL: NCT01415284
Title: ED50 Determination of Hydroxyethylstarch for Treatment of Hypotension During Cesarean Section Under Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Christian Loubert, Dr, Maisonneuve-Rosemont Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LoubertHMR2011/01
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Obstetric Anesthesia; Spinal Anesthesia; Hypotension; Fluid Therapy; Cesarean Section
Keywords: Obstetric anesthesia; Spinal anesthesia; Hypotension; Fluid therapy; Cesarean section; phenylephrine; cardiac output
MeSH Terms: conditions — Hypotension | interventions — HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxyethylstarch 130/0.4 (Experimental)
  Interventions: Drug: Hydroxyethylstarch 130/0.4

INTERVENTIONS:
Drug: Hydroxyethylstarch 130/0.4 — first patient : 500 mL. Following volumes according to up-down sequential allocation, with increments or decrements of 100 mL. An absence of hypotension will lead to an decrement while a presence of hypotension will result in an increment.
  Other Names: Voluven

SUMMARY:
The purpose of this trial is to determine the effective volume of hydroxyethylstarch 130/0.4 which would prevent the occurence of maternal hypotension in 50% of healthy pregnant women undergoing a cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
The incidence of spinal anesthesia-induced hypotension in pregnant women undergoing a cesarean section is high. A preoperative fluid bolus of undetermined volume is frequently administered to lower the incidence of maternal hypotension, with a somewhat poor efficacy. Recently, several investigations have shown that the use of a phenylephrine infusion after the induction of spinal anesthesia results in a significant reduction in hypotensive episodes. Given the high efficacy of this therapy (incidence of hypotension around 20%), it is possible to determine the effective volume of fluid which would prevent hypotension in 50% of the patients studied (ED50).

Healthy term pregnant women undergoing elective cesarean section under spinal anesthesia will be recruited in this trial. The spinal anesthesia regimen will be standardized and all subjects will receive a phenylephrine infusion. The fluid investigated is hydroxyethylstarch (HES) 130/0.4 (Volulyte(R)). The ED50 will be determined using an up-down sequential allocation method initially described by Dixon & Massey. The determination of the HES ED50 will help the anesthesiologist in further treating maternal hypotension appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women (ASA I or II)
* Normal pregnancy
* Term gestation (37 weeks and above)
* Elective cesarean section
* Spinal anesthesia

Exclusion Criteria:

* Cardiopathies
* Hypertensive disease/ pre-eclampsia / eclampsia
* Any contraindication to neuraxial anesthesia
* Patient refusal
* Body mass index > 30 at first antenatal visit and > 32 at cesarean section
* Twin pregnancy
* Known allergies to HES
* Emergency cesarean section

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Volume of HES which will prevent hypotension if 50 % of the subjects. | 4 months

SECONDARY OUTCOMES:
Incidence of hypotension episodes | 1 hour
Incidence of hypertensive episodes | 1 hour
cardiac output | 1 hour
Apgar score | 10 minutes
umbilical artery pH | 2 hours
additional vasopressors administered | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Christian Loubert, MD, FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada